CLINICAL TRIAL: NCT00541281
Title: Randomized Phase Ii Trial Of Weekly Docetaxel, Estramustine And Prednisone Versus Docetaxel And Prednisone In Patient With Hormone-Resistant Prostate Cancer
Brief Title: Safety and Efficacy Study of of Docetaxel vs Docetaxel Estramustine in Hormone Refractory Prostatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL-ONCO 04-001
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Hormone Resistant Prostate Cancer; Metastatic Prostate Cancer
Keywords: prostate cancer; hormone resistant; metastatic; estramustine combine to docetaxel; randomized study
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Docetaxel; Estramustine; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): weekly docetaxel and prednisone
  Interventions: Drug: docetaxel; Drug: estramustine; Drug: prednisone
- B (Active Comparator): weekly docetaxel (35mg/m&) plus prednisone 10mg a day associated with estramustine form day 1to 5 and 8 to 12
  Interventions: Drug: docetaxel; Drug: prednisone

INTERVENTIONS:
Drug: docetaxel — 35mg/m² on day 2 and 9 (21days in a cycle)
  Other Names: Taxotere
Drug: estramustine — 140mg caps x3 bid from day 1to 5 and day 8 to 12 of each cycle
  Other Names: estramustine phosphate
  Arms: A
Drug: prednisone — 2x5 mg a day
  Other Names: medrol

SUMMARY:
we propose to randomize patients with hormone resistant prostate cancer between docetaxel/estramustine/prednisone and docetaxel/prednisone in a phase II study. The principal endpoint will be the efficacy in term of PSA response.

DETAILED DESCRIPTION:
The addition of estramustine to other chemotherapeutic agents that affect microtubule function may improve their efficacy15, 16, 17, 18. A phase III trial compared vinblastine versus the combination of vinblastine plus estramustine as treatment for patients with hormone-refractory prostate cancer. They showed that the association of estramustine and vinblastine was superior to vinblastine alone for time to progression, PSA response and survival (Hudes et al., ASCO 2002). In addition, Berry et al. found that estramustine/paclitaxel improved PSA response rate but not overall survival compared with paclitaxel alone (Berry et al. ASCO2001).

Similar association has been studied with docetaxel. In a phase I trial combining docetaxel and estramustine19, 53% of patients reported a decrease in narcotic use and 63% experienced a PSA response. In another phase I trial, a reduction in PSA of 50% or more was observed in 14 of 17 patients (82%)20. In a phase II trial involving 35 patients, a PSA response was reported in 74% of the patients and objective response in 4 out of 7 patients with measurable disease21. Median survival 22 months in this last study. These studies as well as other support the combination of estramustine and docetaxel in the treatment of HRPC22, 23.

Recently, Oudard et al. competed a phase II randomized study comparing mitoxantrone/prednisone versus docetaxel/estramustine prednisone24. Docetaxel was given either weekly or every 3 weeks. Association of docetaxel/estramustine was found superior to mitoxantrone in term of PSA response, (67-63% versus 18%), clinical benefit (79-56% versus 41%) and survival (19.2 months versus 11.6 months). In addition, toxicities of these regimens were manageable and predictable. In this study, patients received 2 mgr of coumadin to prevent thromboembolic event due to estramustine and only 7 % of the patients had thrombosis. Other grade III & IV toxicities of the estramustine/docetaxel combination included neutropenia (37% in the 3-week regimen and 0 % in the weekly regimen) nausea/vomiting (2% in the 3-week regimen and 0 % in the weekly regimen), diarrhea (7% in the 3-week regimen and 0 % in the weekly regimen). No febrile neutropenia was observed.

Although these data support a role for chemotherapy combinations, such as estramustine and docetaxel, in the treatment of HRPC, further studies are needed to determine the relative contribution of estramustine to the efficacy of docetaxel/estramustine regimen. In this context, we propose to randomize patients with hormone resistant prostate cancer between docetaxel/estramustine/prednisone and docetaxel/prednisone in a phase II study. The principal endpoint will be the efficacy in term of PSA response. We chose to use the weekly regimen as described by Oudard since the toxicity of this regimen is well described and is easily manageable in our experience.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to beginning protocol specific procedures.
* 18 years
* Histologically/cytologically proven prostate adenocarcinoma.
* Documented metastatic prostate adenocarcinoma
* Patients must have received prior hormonal therapy as defined below:
* Castration by orchiectomy and/or LHRH agonists with or without
* Antiandrogens
* Other hormonal agents (e.g., ketoconazole, ...)
* Testosterone level should be < 50 ng/dl in all patients (castrated level).
* Respect of antiandrogen withdrawal period
* No prior chemotherapy regimen at the exception of estramustine phosphate.
* documented disease progression defined either (i) by PSA increase and/or (ii) imaging:
* Prior radiation therapy (to less or equal than 25% of the bone marrow only) is allowed. At least 4 weeks must have elapsed since the completion of radiation therapy and the patient must have recovered from side effects.
* Prior surgery is allowed. At least 4 weeks must have elapsed since the completion of surgery.
* Life expectancy > 3 months.
* ECOG performance status 0-2.
* Normal cardiac function.

Exclusion Criteria:

* Prior chemotherapy except estramustine phosphate.(2)
* Prior isotope therapy
* Prior radiotherapy to >25% of bone marrow
* Prior malignancy except the following: adequately treated basal cell or squamous cell skin cancer, or any other cancer from which the patient has been disease-free for >5 years.
* Known brain or leptomeningeal involvement.
* Symptomatic peripheral neuropathy > grade 2
* Other serious illness or medical condition
* Concurrent treatment with other experimental drugs.
* Treatment with any other anti-cancer therapy (except LHRH agonists)
* Treatment with systemic corticosteroids used for reasons other than specified by the protocol must be stopped prior to the administration of docetaxel.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-12; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of the association of Docetaxel and Estramustineand Prednisone versus Docetaxel and Prednisone in the treatment of hormone refractory prostate cancer in terms o PSA response | within 30 days after end of treatment

SECONDARY OUTCOMES:
PSA response Time to PSA progression PSA response duration Event Progression-Free Survival Overall survival Palliative response (Pain) Safety Objective response measurable disease (RECIST) | untill death occurs

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, MD PHD, Principal Investigator — Cliniques Universitaires St Luc; Joseph Kerger, MD, Principal Investigator — Clinqiue Universitaire de Mont Godinne
Locations (19):
- Belgium (18):
  - St Pierre, Ottignies, Brabant Wallon
  - Notre Dame et Reine Fabiola, Charleroi, Hainaut
  - RHMS louis caty, Baudour
  - Clinique Saint Luc, Bouge
  - CHR Warquignies, Boussu
  - Az klina, Brasschaat
  - Parc Léopold, Brussels
  - Hôpitaux IRIS Sud, Brussels
  - Cliniques Universitaires St luc, Brussels
  - Sint Nilolaus, Eupen
  - Clinique St Joseph, Gilly
  - Notre Dame de Grâce, Gosselies
  - CH Jolimont Lobbes, La Louvière
  - St Joseph, Liège
  - CHU Ambroise paré, Mons
  - clinique Sainte Elisabeth, Namur
  - Notre Dame, Tournai
  - Clinique Universitaire de Mt Godinne, Yvoir
- CHR Luxembourg, Luxembourg, Luxembourg